CLINICAL TRIAL: NCT07068425
Title: Retrospective and Prospective Longitudinal Observational Study on Immune Thrombocytopenia
Brief Title: Longitudinal Observational Study on Immune Thrombocytopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology Affiliation: Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: PKU-ITP2025
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective cohort: Patients whose first visit to our institution and the termination of follow-up both occurred before the opening of this study will contribute to the retrospective cohort.
- Prospective cohort: Patients whose first visit to our institution occur after the opening of this study will contribute to the prospective cohort.
- Retrospective/Prospective cohort: Patients whose first visit to our institution occurred before the opening of this study and whose follow-up will terminate after the opening of this study will contribute to the ambispective cohort.

SUMMARY:
Immune Thrombocytopenia (ITP) is a bleeding disorder characterized by immune-mediated destruction and/or impaired production of platelets, leading to clinical manifestations such as petechiae, purpura, mucosal bleeding, and in severe cases, life-threatening visceral or intracranial hemorrhage. Research on the diagnosis, treatment, and prognosis of ITP is critical for improving patient outcomes and quality of life. However, most existing hematologic cohort studies are limited to single-center or small multicenter samples, lacking comprehensive, large-scale prospective investigations.

To address this gap, our center plans to conduct a large-sample, combined retrospective and prospective longitudinal observational cohort study of ITP patients. The study will enroll patients to collect baseline demographic and diagnostic data, followed by longitudinal follow-up via questionnaires, telephone interviews, video consultations, online platforms, and in-person visits. Key variables including treatment regimens, comorbidities, and prognostic outcomes will be systematically recorded. Additionally, hospitalization and outpatient expenditure data will be extracted from electronic medical records.

This study aims to provide high-quality real-world evidence on the epidemiology, treatment patterns, clinical outcomes, and healthcare costs of ITP patients in China, ultimately informing clinical decision-making and health policy.

DETAILED DESCRIPTION:
Immune Thrombocytopenia (ITP) is an immune-mediated acquired bleeding disorder characterized by thrombocytopenia with normal or increased megakaryocytes in the bone marrow accompanied by maturation defects. Epidemiological studies estimate its incidence at approximately 2-5 cases per 100,000 individuals in the general population.

The primary clinical manifestation of ITP is bleeding, ranging from minor cutaneous/mucosal hemorrhage to life-threatening organ bleeding. Notably, some patients also exhibit increased risk of thrombotic/embolic events. Embolic complications in critical organs (e.g., heart, brain) may significantly impair quality of life and lead to life-threatening conditions.

Currently, most ITP cohort studies in China are limited to single-center designs or small multicenter studies with insufficient sample sizes. There remains a notable lack of large-scale, longitudinal prospective cohort studies.

To address these limitations, this multicenter, retrospective-prospective longitudinal observational study will enroll diagnosed ITP patients to systematically collect:

Baseline demographic and diagnostic data Prospective follow-up data via questionnaires, telemedicine, and clinical visits Treatment regimens, comorbidities, and prognostic outcomes Healthcare utilization costs through electronic medical records

By establishing this comprehensive real-world database, the study aims to:

Elucidate the epidemiology, treatment patterns, and economic burden of ITP in China Provide evidence-based support for developing novel clinical strategies Improve long-term hemorrhage-free survival rates This investigation will serve as a foundational platform for optimizing ITP management and enhancing patient outcomes across China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of ITP
2. Patients treated at Peking University People's Hospital since January 1, 2005

Exclusion Criteria:

1. Any condition that may render follow-up data unreliable, including but not limited to severe psychiatric disorders"
2. Patients deemed ineligible for the study by investigators"

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed immune thrombocytopenia (ITP).
  Diagnostic Criteria for ITP:
  1. Sustained platelet count <100×10⁹/L
  2. Normal or increased megakaryocyte count in bone marrow with maturation defects
  3. Exclusion of other potential causes of thrombocytopenia including: pseudothrombocytopenia, drug-induced thrombocytopenia, viral infections, helicobacter pylori infection, hematologic disorders, autoimmune diseases, hypersplenism, malignancies
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis | 5 years
  To analyze the long-term prognosis of patients with immune thrombocytopenia (ITP), and analyze the risk factors associated with their prognosis.
Overall response rate | 180 days
  To analyze the therapeutic efficacy of patients with ITP, and analyze the impact factors associated with the efficacy.
Long-term overall remission rate | 1 year
  Proportion of the participants with an overall remission.
Comorbidities | 5 years
  The incidence, risk factors, treatments, and prognosis of complications

SECONDARY OUTCOMES:
Incidence | 5 years
  To describe the incidence of ITP, and analyze the risk factors associated with these diseases.
Safety of treatment | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Health economic evaluation | 5 years
  To perform hospital stay and hospitalization cost evaluation in patients with thrombosis and hemostasis diseases

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing 100010, Beijing, China